CLINICAL TRIAL: NCT02318316
Title: "Exhaled Breath Condensate" in Allogeneic Stem Cell Recipients and Value in Follow-up
Brief Title: "Exhaled Breath Condensate" in Allogeneic Stem Cell Recipients and the Value in Follow-up
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nilgün Yılmaz Demirci, MD, Gazi University
Other Study IDs: EBC01
Record Dates: First submitted 2014-12-10; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Exhaled Breath Condensate
Keywords: Exhaled breath condensate; allogeneic stem cell transplantation; pulmonary complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EBC level: Exhaled breath condensate level of allogeneic stem cell transplantation patients
  Interventions: Other: Exhaled breath condensate

INTERVENTIONS:
Other: Exhaled breath condensate — Breath condensate samples will be collected with a commercially available condenser (EcoScreen®, Erich Jaeger, Germany). Subjects will breathe through a mouthpiece and a two-way non-rebreathing value in which inspiratory and expiratory air were separated, and saliva was trapped. They will be asked to breathe at a normal frequency and tidal volume for 15 minutes while wearing nose clips, allowing collection of 1.5-2.5 mL of condensate. After collecting this, pH will be measured and the waste collection will be stored at -80 degrees. Then 8 isoprostane and nitrotyrosine will be measured collectively

SUMMARY:
The most effective treatment of hematologic malignancies and some benign hematological diseases is allogeneic stem cell transplantation therapy. Pulmonary complications can occur after allogeneic stem cell transplantation. And these complications effect mortality and morbidity in these patients. In this study we want to investigate the use of exhaled breath condensate (EBC) collection which is a simple and completely noninvasive method. By this way we hope to detect pulmonary complications early. EBC, has been implicated in the pathophysiology of inflammatory airway diseases such as cystic fibrosis, asthma, chronic obstructive pulmonary disease (COPD) and bronchiectasis. EBC, has not been investigated before in patients who underwent stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* hematologic malignancies or benign hematological diseases that allogeneic stem cell transplantation performed

Exclusion Criteria:

* allogeneic stem cell transplantation patients with Asthma or COPD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: allogeneic stem cell transplantation patients for hematologic malignancies and some benign hematological diseases
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The pH level of exhaled breath condansate | 2 years

SECONDARY OUTCOMES:
The nitrotyrosine and 8-isoprostane levels of exhaled breath condansate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Yıldırım, professor, Principal Investigator — Gazi University Faculty of Medicine Chest Disease Department

REFERENCES:
- [Background] Horvath I, Hunt J, Barnes PJ, Alving K, Antczak A, Baraldi E, Becher G, van Beurden WJ, Corradi M, Dekhuijzen R, Dweik RA, Dwyer T, Effros R, Erzurum S, Gaston B, Gessner C, Greening A, Ho LP, Hohlfeld J, Jobsis Q, Laskowski D, Loukides S, Marlin D, Montuschi P, Olin AC, Redington AE, Reinhold P, van Rensen EL, Rubinstein I, Silkoff P, Toren K, Vass G, Vogelberg C, Wirtz H; ATS/ERS Task Force on Exhaled Breath Condensate. Exhaled breath condensate: methodological recommendations and unresolved questions. Eur Respir J. 2005 Sep;26(3):523-48. doi: 10.1183/09031936.05.00029705. PMID 16135737
- [Background] Dupont LJ, Dewandeleer Y, Vanaudenaerde BM, Van Raemdonck DE, Verleden GM. The pH of exhaled breath condensate of patients with allograft rejection after lung transplantation. Am J Transplant. 2006 Jun;6(6):1486-92. doi: 10.1111/j.1600-6143.2006.01331.x. PMID 16686775
- [Background] Mo XD, Xu LP, Liu DH, Zhang XH, Chen H, Chen YH, Han W, Wang Y, Wang FR, Wang JZ, Liu KY, Huang XJ. Risk factors for bronchiolitis obliterans syndrome in allogeneic hematopoietic stem cell transplantation. Chin Med J (Engl). 2013 Jul;126(13):2489-94. PMID 23823823